CLINICAL TRIAL: NCT02892552
Title: Cone Beam CT Versus Multislice CT: Radiologic Diagnostic Agreement in the Postoperative Assessment of Cochlear Implantation
Brief Title: Cone Beam CT Versus Multislice CT in the Postoperative Assessment of Cochlear Implantation
Acronym: COCOBE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012.736
Record Dates: First submitted 2016-09-02; First posted 2016-09-08 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2016-08

CONDITIONS: Cochlear Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cone Beam (Experimental): Patients included will have first a MultiSlice Computed tomography (MSCT) as usual and then a Cone Beam Computed Tomography (CBCT)
  Interventions: Radiation: Cone Beam Computed Tomography (CBCT); Radiation: Multiple Detector Computed Tomography (MDCT)

INTERVENTIONS:
Radiation: Cone Beam Computed Tomography (CBCT) — Patients had an additional Cone Beam Computed Tomography, after the usual MDCT
Radiation: Multiple Detector Computed Tomography (MDCT) — Patients had a usual MDCT, before having an additional Cone Beam Computed Tomography

SUMMARY:
Objective: To evaluate the diagnostic concordance between multislice computed tomography (MSCT) and cone beam computed tomography (CBCT) in the early postoperative assessment of patients after cochlear implantation.

Study Design: Prospective, randomized, single-center, interventional, pilot study on the diagnostic performance of a medical device.

Setting: Tertiary referral center. Patients: Patients aged over 18 years requiring a CT scan after cochlear implant surgery.

Interventions: Nine patients were implanted with electrode arrays from three different manufacturers, including one bilateral. High-resolution MSCT and CBCT were then performed, and 2 experienced radiologists blinded to the imaging modality evaluated the randomized images, twice.

ELIGIBILITY:
Inclusion Criteria:

* CI surgery for severe to profound bilateral deafness
* affiliated with the French health insurance

Exclusion Criteria:

* pregnancy
* Patients weighing more than 160 kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Concordance between MDCT and CBCT for assessing the scalar position of the electrodes | At inclusion
  Blinded images were analyzed in random order by 2 radiologists with several years of experience in temporal bone imaging. Each radiologist analyzed on the workstation the images of each patient twice at 4- to 8-week intervals. A consensus reading was performed by a third experienced radiologist in case of discordance.
  Each radiologist determined CI localization. The cochlear implant (CI) was considered within the scala tympani if it was in the most posterior scala on axial reconstructions passing through the cochlea (behind the osseous spiral lamina often seen).

SECONDARY OUTCOMES:
length of the intracochlear electrode array | At inclusion
  Blinded images were analyzed in random order by 2 radiologists with several years of experience in temporal bone imaging. Each radiologist analyzed on the workstation the images of each patient twice at 4- to 8-week intervals. A consensus reading was performed by a third experienced radiologist in case of discordance.
  This measurement was performed in the oblique coronal plane of the cochlea.
percentage of implanted cochlea | At inclusion
  Blinded images were analyzed in random order by 2 radiologists with several years of experience in temporal bone imaging. Each radiologist analyzed on the workstation the images of each patient twice at 4- to 8-week intervals. A consensus reading was performed by a third experienced radiologist in case of discordance.
  This measurement was performed in the oblique coronal plane of the cochlea.
number of intracochlear electrodes | At inclusion
  Blinded images were analyzed in random order by 2 radiologists with several years of experience in temporal bone imaging. Each radiologist analyzed on the workstation the images of each patient twice at 4- to 8-week intervals. A consensus reading was performed by a third experienced radiologist in case of discordance.
  This measurement was performed in the oblique coronal plane of the cochlea.
radiation dose | At inclusion
  Radiation dose was estimated using Computed Tomography Dose Index (CTDI, in Gy.cm) for each patient and scanner. These data are collected directly from the data sheet for each examination (also anonymised).

CONTACTS AND LOCATIONS:
Locations (1):
- Service imagerie pavillon B, Hopital E. Herriot, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Razafindranaly V, Truy E, Pialat JB, Martinon A, Bourhis M, Boublay N, Faure F, Ltaief-Boudrigua A. Cone Beam CT Versus Multislice CT: Radiologic Diagnostic Agreement in the Postoperative Assessment of Cochlear Implantation. Otol Neurotol. 2016 Oct;37(9):1246-54. doi: 10.1097/MAO.0000000000001165. PMID 27518208